CLINICAL TRIAL: NCT01749085
Title: A Phase 1, Open Label Study In Healthy Subjects To Estimate The Effect Of Food And The Drug-Drug Interaction Potential Of Ketoconazole On PF-04449913 Pharmacokinetics
Brief Title: Study To Determine The Effect Of Food And Strong CYP3A4 Enzyme Inhibitor On PF-04449913 Drug Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1371010
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Healthy Volunteers
Keywords: PF-04449913; Food Effect; Drug-drug interaction; CYP3A4 inhibitor; Pharmacokinetics
MeSH Terms: interventions — glasdegib; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental)
  Interventions: Drug: PF-04449913, ketoconazole
- Sequence 2 (Experimental)
  Interventions: Drug: PF-04449913, ketoconazole

INTERVENTIONS:
Drug: PF-04449913, ketoconazole — Subjects receive a 200 mg oral dose of PF-04449913 under fasted conditions with washout, then single 200 mg oral dose of PF-04449913 under fed with washout and finally a single 200 mg dose 0f PF-04449913 following dosing to steady state with ketoconazole
  Arms: Sequence 1
Drug: PF-04449913, ketoconazole — Subjects receive a 200 mg oral dose of PF-04449913 under fed conditions with washout, then single 200 mg oral dose of PF-04449913 under fasted with washout and finally a single 200 mg dose of PF-04449913 following dosing to steady state with ketoconazole
  Arms: Sequence 2

SUMMARY:
The study aims to determine what effect a high fat meal will have on the drug exposure of PF-04449913. The study also aims to determine the effect of a strong enzyme (CYP3A4) inhibitor on drug exposure of PF-04449913.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 and 55 years (inclusive):Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen
* 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at Screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility. Subjects with one of the following currently in the past 6 months: myocardial infarction, congenital long QT syndrome, torsades de pointes or clinically significant ventricular arrhythmias.
* Pregnant or nursing females and females of childbearing potential including those with tubal ligation. To be considered for enrollment, women of 45 to 55 years of age who are postmenopausal (defined as being amenorrheic for at least 2 years) must have confirmatory FSH test results at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 8 days
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 8 days

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 8 days
Apparent Oral Clearance (CL/F) | 8 days
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 8 days
Apparent Volume of Distribution (Vz/F) | 8 days
Plasma Decay Half-Life (t1/2) | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371010&StudyName=Study%20To%20Determine%20The%20Effect%20Of%20Food%20And%20Strong%20CYP3A4%20Enzyme%20Inhibitor%20On%20PF-04449913%20Drug%20Levels